CLINICAL TRIAL: NCT07250061
Title: Augmenting Cognitive Processing Therapy With a Peer Led Support Intervention to Improve Well-Being: A Sustainable and Scalable Model for Enhancing PTSD Recovery in Vulnerable Populations
Brief Title: Self-Help Cognitive Processing Therapy (CPT)/Women Veterans Network (WoVeN) Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-46292; 1R34MH138605-01A1 (NIH)
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Posttraumatic Stress Disorder; Depression
Keywords: Mental well being; Self help cognitive processing therapy; Peer support program; Quality of life; Loneliness; Women Veterans Network
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Psychological Well-Being | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: A three-arm, randomized, controlled clinical trial will be conducted with a national sample of women veterans who suffer from PTSD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self-Help Cognitive Processing Therapy (shCPT) (Experimental): Participants randomized to this arm will receive Cognitive Processing Therapy (CPT) and a self- help book.
  Interventions: Behavioral: Self-Help Cognitive Processing Therapy
- Women Veterans Network (WoVeN) + self-help CPT (BOTH) (Experimental): Participants randomized to this arm will receive Cognitive Processing Therapy by trained peer leaders from the Women Veterans Network (WoVeN).
  Interventions: Behavioral: Self-Help Cognitive Processing Therapy; Behavioral: Women Veterans Network (WoVeN)
- Treatment as Usual (TAU) (Active Comparator): Participants randomized to this arm will receive TAU.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Self-Help Cognitive Processing Therapy — Participants will be given a copy of the CPT self-help book that guides the trauma survivor through the same CPT protocol that is typically delivered by a therapist but supplemented with significant additional guidance and suggestions to aid the survivor in their journey toward recovery. This 10-week program also provides links to educational videos, fillable worksheets, and resources for the individual if they would like to seek additional care
  Other Names: shCPT
  Arms: Self-Help Cognitive Processing Therapy (shCPT); Women Veterans Network (WoVeN) + self-help CPT (BOTH)
Behavioral: Women Veterans Network (WoVeN) — Participants will complete the CPT self-help book while also enrolled in a WoVeN group. WoVeN is a national, peer support network with groups led by women veterans, for women veterans. During this 8-week program, Peer Leaders who are trained by national experts in the WoVeN curriculum conduct weekly groups. Groups consist of approximately 4-8 women veterans, each lasting about 90 minutes, and focus on relevant themes such as life transitions, balance, hope, connections, trust, and esteem.
  Other Names: BOTH
  Arms: Women Veterans Network (WoVeN) + self-help CPT (BOTH)
Other: Treatment as Usual — Participants will receive psychoeducation about PTSD and different treatment options using the materials developed by the VA National Center for PTSD. They will also be provided with a referral list with guidance and suggestions and assistance in navigating the list and the referral process. All interventions must be completed within 10 weeks.
  Other Names: TAU
  Arms: Treatment as Usual (TAU)

SUMMARY:
Posttraumatic stress disorder (PTSD) can have significant impairment on aspects of mental well-being (MWB) including functioning, loneliness, physical health, and quality of life. There are several evidence-based treatments (EBPs) effective in treating PTSD such as Cognitive Processing Therapy (CPT) which is a specific type of cognitive behavioral therapy that has been proven effective in reducing symptoms of PTSD. However, there are several barriers (e.g., lack of providers, waitlists, costs, stigma, disabilities that complicate travel) that can prevent someone from engaging with these treatments. Recently, a self-help version of CPT was created to help address these barriers; but little research has been conducted to test its efficacy. Further, less is know about how a peer support program may augment improvements from participating in an EBP. The Women Veteran Network (WoVeN), a peer support program designed for women veterans, has a manualized 8-week program that directly targets MWB. It has been found to help foster belongingness and connectedness, particularly in those suffering from PTSD and depression.

The present study aims to establish the feasibility, acceptability and tolerability of a scalable, sustainable, and effective treatment option for trauma survivors with subthreshold or full PTSD. The overarching goal is to understand the effectiveness of a self-help version of an EBP (either alone or in combination with a peer support program) in reducing PTSD symptoms while also helping improve mental well-being, reduce barriers, and increase access to quality care within health disparity populations.

DETAILED DESCRIPTION:
The design for this study is a three-arm, randomized, controlled clinical trial (RCT) with a national sample of women veterans who suffer from PTSD. Participants will be recruited from WoVeN and from the women veteran population. Treatment conditions will be 1.) self-help CPT only (shCPT), 2.) concurrent WoVeN + self-help CPT (BOTH), or 3.) referral + treatment as usual (TAU). All treatments must be completed within 10 weeks. Ninety women will be randomized in a 1:1:1 ratio across the three treatment conditions. Patient participants will be asked to complete three major assessments (baseline, post-treatment, three month follow up) that consist of a structured interview and questionnaire. These major assessment will take ~2.5 hours to complete. Participants will also be asked to complete weekly surveys that will help monitor ongoing progress engagement with the intervention. Before the RCT launches, an open trial involving 6 women will pilot the BOTH condition. Information gathered from this will be used to refine the study before recruiting more women.

ELIGIBILITY:
Inclusion Criteria:

* Identifies as a woman
* Has served in the United States military
* A full or subthreshold (meets criteria for 2 out of 4 of the symptom clusters for PTSD) Post Traumatic Stress Disorder (PTSD) diagnosis
* Able to read English well enough to complete study questionnaires

Exclusion Criteria:

* Clinician judgment that the participant is not appropriate for self-help level of care for PTSD (i.e., recent psychiatric hospitalization, requires detox, volatile, active suicidality)
* Current psychosis or unstable bipolar disorder (determined during baseline interview as described in screening and enrollment procedures)
* Must not have participated in a WoVeN group within the last year
* Must not be receiving an evidenced-based therapy for PTSD at the time of the screening

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Clinician assessed PTSD Symptoms | Pre intervention- baseline, Post intervention- 10 weeks, Follow-up- 28 weeks
  This outcome will be assessed with the Clinician-Administered PTSD Scale for the Diagnostic and Statistical Manual of Mental Illnesses (DSM-5) (CAPS-5). It obtains information about frequency and intensity for the 20 PTSD symptoms using a 5-point ordinal scale from 0 (absent) to 4 (extreme/incapacitating), based on the patient's frequency and intensity of the symptom. The final score is a total severity score that can range from 0 to 80 with higher scores indicating more severe PTSD symptoms.

SECONDARY OUTCOMES:
Self reported depression | Pre intervention- baseline, Post intervention- 10 weeks, Follow-up- 28 weeks
  This outcome will be assessed with the Patient Health Questionnaire-9 (PHQ-9) which is a a 9-item brief assessment of current depressive symptoms using a 4-point Likert scale from 0 (not at all) to 3 (nearly every day). The final score is a total severity score that can range from 0 to 27 with higher scores indicating more severe depression symptoms.
Mental well being | Pre intervention- baseline, Post intervention- 10 weeks, Follow-up- 28 weeks
  This outcome will be assessed with the Ryff's Psychological Well-Being Scale which is a 42 item self-report assessment that measures 6 aspects of well-being and happiness including autonomy, environmental mastery, personal growth, positive relationships with others, purpose in life, and self-acceptance on a Likert scale from 1 (strongly agree) to 7 (strongly disagree). A higher score on a subscale indicates a greater degree of well-being in that area.
Self reported PTSD | Pre intervention- baseline, Post intervention- 10 weeks, Follow-up- 28 weeks
  This outcome will be assessed with the PTSD Checklist -DSM-5 (PCL-5), a 20-item assessment of the respondent's reactions to a potentially traumatic experience, according to the DSM-5 symptom criteria for PTSD. The PCL-5 uses a 5-point Likert scale from 0 (not at all) to 4 (extremely). This results in a total symptom severity score ranging from 0 to 80, with higher scores indicating more severe symptoms.
Belongingness | Pre intervention- baseline, Post intervention- 10 weeks, Follow-up- 28 weeks
  This outcome will be assessed with the The General Belongingness Scale (GBS) a 12-item scale that assesses general feelings of belonging on a Likert scale of 1= strongly disagree to 7= strongly agree. Six items are included on the acceptance/inclusion subscale and the other six load onto the rejection/exclusion subscale. The total score ranges from 12 to 84, with higher scores indicating a greater sense of belonging
Trauma Related Cognitions | Pre intervention- baseline, Post intervention- 10 weeks, Follow-up- 28 weeks
  This outcome will be assessed with the Posttraumatic Cognitions Inventory - 9 item (PTCI-9) which is a 33 item assessment of trauma-related thoughts and beliefs. The assessment yields 3 subscales, negative thoughts of self, negative thoughts about the world, and self-blame. Higher total scores and subscale scores indicate a greater endorsement of negative post-traumatic cognitions.

CONTACTS AND LOCATIONS:
Overall Officials: Tara E Galovski, PhD, Principal Investigator — BUCA School of Medicine, Psychiatry and VA Medical Center

IPD SHARING:
Plan to Share IPD: No